CLINICAL TRIAL: NCT03321812
Title: Clinical Study of Decalcification Bone Scaffold for Cartilage Lesions of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Ao Yingfang, Director of the Institute of Sports Medicine , Principal Investigator, Clinical Professor of Orthopedic Sports Medicine, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-AO-01
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Cartilage Injury
Keywords: decalcification bone scaffold; microfracture; randomized controlled trial; cartilage lesions of the knee
MeSH Terms: conditions — Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- decalcification bone scaffold (Experimental): Decalcification bone scaffold is a novel tissue engineered acellular matrix scaffold with the closest biomechanics and structure to normal cartilage.
  Interventions: Procedure: decalcification bone scaffold; Procedure: microfracture
- Microfracture (Active Comparator): Microfracture is a conventional treatment for cartilage lesions of the knee.
  Interventions: Procedure: microfracture

INTERVENTIONS:
Procedure: decalcification bone scaffold — Decalcification bone scaffold is a tissue engineering acellular matrix scaffold with the closest biomechanics and structure of normal cartilage.
  Arms: decalcification bone scaffold
Procedure: microfracture — Microfracture is the surgical option for conventional treatment of cartilage defects.

SUMMARY:
The trial evaluates the clinical efficacy and safety of decalcification bone scaffold for cartilage lesions of the knee. Half of participants will receive decalcification bone scaffold combined with microfracture, while the other will only receive microfracture as a control group.

DETAILED DESCRIPTION:
Decalcification bone scaffold is a tissue engineering scaffold with the closest biomechanics and structure of normal cartilage. The objective of the study is to evaluate the clinical efficacy of arthroscopic decalcification bone scaffold combined with microfracture in the repairment of articular cartilage defects by randomized controlled trial. Sixty patients with clinically diagnosed knee cartilage injury according to 1: 1 were divided into experimental group and control group. The experimental group will be treated with decalcification bone scaffold combined with microfracture .The control group will be treated with microfracture . The patients will be treated by the same surgeon in this study group. MRI evaluation, Lysholm score, IKDC score, Tegner score, VAS score are selected as the measures of outcome, while the blood routine, blood biochemistry, urine, CRP, ECG and other laboratory tests will be recorded inclduing the incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old, male or female
* Cartilage defect 2-8 cm²
* Subjects have the surgical indication of microfracture and no contradiction
* Subjects participate the clinical trial voluntarily, and sign informed consent
* Subjects could comply with follow-up

Exclusion Criteria:

* Participated in other drug or medical device clinical trials in the last 6 months.
* Can not accept allogeneic decalcified bone due to religion, ethnic and other issues.
* Defect area 2 cm² or 8 cm² or lack of normal cartilage tissue around defect zone.
* Complex multi-ligament injury
* Suffered from systemic immune disease or systemic, locally infected
* Joint fibrosis, joint rigidity, mobility was significantly limited
* Moderate and severe osteoarthritis
* With contraindications to MRI
* Hemophilia
* General condition can not tolerate surgery
* Pregnant or planned pregnant women and lactating women
* With abnormal spirit and selfless ability
* Other circumstances judged by doctors that can not participate in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Appraise of magnetic reasonance imaging | 5 years
  Evaluate the articular cartilage postoperatively by MRI.

SECONDARY OUTCOMES:
Lysholm score | 5 years
  The Lysholm score consists of eight items including limping, locking, pain, stair climbing, use of supports, instability, swelling, and squatting. The higher values represent a better outcome.
International Knee Documentation Committee (IKDC) 2000 | 5 years
  International Knee Documentation Committee (IKDC) 2000. The higher values represent a better outcome.
Tegner activity level score | 5 years
  The highest level of activity that you participated in before your injury and the highest level you are able to participate in currently. The higher values represent a better outcome.
Visual analogue scale | 5 years
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. From 0 to 10, no pain 0, worst pain imaginable 10. The higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yingfang Ao, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No